CLINICAL TRIAL: NCT05282940
Title: Bioavailability of a Formulation of Levonorgestrel and Ethinyl Estradiol 15.0 mg/0.03 mg Coated Tablets With Regards to the Marketed Reference Product
Brief Title: Bioavailability of Levonorgestrel and Ethinyl Estradiol Tablets 15.0 mg/0.03 mg With Regards to Reference Product
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Andromaco S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HP8814-03
Record Dates: First submitted 2022-02-25; First posted 2022-03-16 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-04

CONDITIONS: Therapeutic Equivalency
MeSH Terms: interventions — Levonorgestrel; Ethinyl Estradiol; Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levonorgestrel and Ethinyl estradiol Test Product (Experimental): Participants will receive two tablets of the test formulation containing Levonorgestrel 15.0 mg and Ethinyl estradiol 0.03 mg. The tablets will be taken with water.
  Interventions: Drug: Levonorgestrel 15.0 mg and Ethinyl estradiol 0.03 mg Test Drug
- Levonorgestrel and Ethinyl estradiol Reference Product (Active Comparator): Participants will receive two tablets of the test marketed reference formulation containing Levonorgestrel 15.0 mg and Ethinyl estradiol 0.03 mg. The tablets will be taken with water.
  Interventions: Drug: Microgynon CD

INTERVENTIONS:
Drug: Levonorgestrel 15.0 mg and Ethinyl estradiol 0.03 mg Test Drug — Investigational Medicinal Product
  Arms: Levonorgestrel and Ethinyl estradiol Test Product
Drug: Microgynon CD — Microgynon CD will be used as a comparator drug for the BE study. Other Name: Levonorgestrel 15.0 mg and Ethinyl estradiol 0.03 mg Reference Drug
  Arms: Levonorgestrel and Ethinyl estradiol Reference Product

SUMMARY:
This study will investigate the bioavailability in women of 2 tablet formulations containing Levonorgestrel 15.0 mg and Ethinyl estradiol 0.03 mg. The study will be performed at a single site with 36 subjects. Participants will take 2 tablets of the test product and reference product in 2 periods and 2 sequences (either test after reference or reference after test). There will be a washout of at least 14 days between each study period.

DETAILED DESCRIPTION:
The primary objective of the study is to investigate the relative bioavailability of Levonorgestrel and Ethinyl estradiol of 2 tablet formulations with Levonorgestrel 15.0 mg and Ethinyl estradiol 0.03 mg and to demonstrate bioequivalence of both formulations in terms of rate and extent of absorption:

* Test Product: Product manufactured by Laboratorios Andrómaco S.A.
* Reference Product: Microgynon [Trademark], product of Bayer AG, Brasil. The 90% confidence intervals for the intra-subject coefficient of variation (Test versus Reference Product) for the main pharmacokinetic parameters área under the plasma concentration-time curve from time zero to time t (AUC0-t) and from time zero to infinite (AUC0-∞), and maximum plasma concentration (Cmax) for total Levonorgestrel and Ethinyl estradiol will be determined. Participants will be confined in the study site for approximately 34 hours during each study period (for 10 hours pre-dosing and for 24 hours post dosing) during which pharmacokinetic (PK) blood samples will be obtained. 21 blood samples will be taken up to 24 hours after the administration in each period. Participants will return to the site to provide additional blood samples at 48 h, and 72 h postdose. The washout period between the two study periods will be at least 14 days. A validated LC-MS/MS bio-analytical method will be used for estimation of plasma levels of Ethinyl-estradiol and Levonorgestrel. The safety objective is to evaluate the tolerability of both formulations in women by collecting adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy non-pregnant, non-breast feeding female literate volunteers of 18 to 45 years (both years inclusive) with BMI of 18.50 - 29.99 Kg/m2 and weight > 50 Kg.
2. Healthy volunteers as evaluated by medical history, vitals and general clinical examination.
3. Normal or clinically insignificant biochemical, hematological, urine and serology parameters.
4. Normal or clinically insignificant EC.
5. Negative urine test for drugs of abuse, negative pregnancy test and do not plan to become pregnant during course of the study and for 03 months after completion of study.
6. Volunteers who are willing to use acceptable methods of contraception (barrier method/IUD/surgical) or abstinence, for the entire duration of the study and do not plan to be pregnant for at least 1 month after the last drug administration.
7. Volunteers who can give written informed consent and communicate effectively.

Exclusion Criteria:

1. History of any major surgical procedure in the past 03 months.
2. History of any clinically significant cardiac, gastrointestinal, respiratory, hepatic, renal, endocrine, neurological, metabolic, psychiatric and hematological disorders.
3. History of chronic alcoholism/ chronic smoking/ drug of abuse.
4. Volunteers with known hypersensitivity to Ethinyl-estradiol and Levonorgestrel or any of the excipients.
5. History of consumption of tobacco containing products within 48 hours prior to proposed time of dosing
6. Volunteer who are positive for hepatitis B surface antigen, anti-hepatitis C antibody, treponemal antibodies and human immunodeficiency virus (HIV 1&2) antibodies.
7. Present or past history of intake of drugs or any prescription drug or over the counter (OTC) drugs within 14 days which potentially modify kinetics / dynamics of Ethinyl-estradiol and Levonorgestrel or any other medication judged to be clinically significant by the investigator.
8. History of consumption of grapefruit and/or its products within 10 days prior to the start of study.
9. Volunteer who had participated in any other clinical study or who had bled during the last 03 months before check-in.
10. History of consumption of one or more of the below, 48 hours prior to dosing: Xanthine containing food or drinks such as cola, chocolate, coffee or tea, citrus fruits or items (lime, lemon and orange), alcohol and any other food/beverage known to have interactions as deemed by the investigator.
11. Volunteers who are dysphagic

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-02-26 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Total Ethinyl estradiol: area under the plasma concentration-time curve from 0 to 72 hours (AUC0-72) | From tablet intake and up to 72 hours after tablet intake
  21 samples up to 72 hours will be taken after the administration in each period
Total Levonorgestrel: area under the plasma concentration-time curve from 0 to 72 hours (AUC0-72) | From tablet intake and up to 72 hours after tablet intake
  21 samples up to 72 hours will be taken after the administration in each period
Total Ethinyl estradiol: Maximum plasma concentration (Cmax) | From tablet intake and up to 72 hours after tablet intake
  21 samples up to 72 hours will be taken after the administration in each period
Total Levonorgestrel: Maximum plasma concentration (Cmax) | From tablet intake and up to 72 hours after tablet intake
  21 samples up to 72 hours will be taken after the administration in each period
Total Ethinyl estradiol: Time to achieve maximum plasma concentration (tmax) | From tablet intake and up to 72 hours after tablet intake
  21 samples up to 72 hours will be taken after the administration in each period
Total Levonorgestrel: Time to achieve maximum plasma concentration (tmax) | From tablet intake and up to 72 hours after tablet intake
  21 samples up to 72 hours will be taken after the administration in each period

CONTACTS AND LOCATIONS:
Locations (1):
- Azidus Laboratories Ltd., Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No